CLINICAL TRIAL: NCT03693040
Title: Digital Health Feedback System (DHFS) for Longitudinal Monitoring of ARVs Used in HIV Pre-exposure Prophylaxis (PrEP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Gilead Sciences (Industry); Proteus Digital Health, Inc. (Industry)
Responsible Party: Principal Investigator, Sara H. Browne, MD, MPH, Principal Investigator, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 161618; R01MH110057 (NIH)
Record Dates: First submitted 2018-07-31; First posted 2018-10-02 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: HIV Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DHFS with IS-Truvada (Experimental): Digital Health Feedback System (DHFS) with IS-Truvada 1 capsule daily for 12 weeks
  Interventions: Device: Digital Health Feedback System

INTERVENTIONS:
Device: Digital Health Feedback System — This intervention uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new technologies approved by the FDA, to collect information about patients taking their PrEP medication. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which provides information about when patients have taken their PrEP medication.

SUMMARY:
This study uses an ingestion sensor and a wearable sensor (worn as a patch on the skin), which are new Proteus Digital Health (PDH) technologies approved by the FDA, to collect information about patients taking their Pre-Exposure Prophylaxis (PrEP) medication for HIV prevention. The wearable sensor records information, which is uploaded wirelessly to a mobile device and then to a secure computer. Together the sensors and the mobile device transmitting the information to the study computer are called a digital health feedback system (DHFS), which gives healthcare providers information about when patients have taken their PrEP medication.

The purpose of the study is to demonstrate that the DHFS is easy to use and acceptable to people taking PrEP; that patients will persist with its use; and that the system provides valid, accurate measures of adherence.

DETAILED DESCRIPTION:
This study is a prospective single arm open label intervention study over 12 weeks using the DHFS with participants initiating or continuing HIV PrEP. The study intervention has an initiation (Phase 1), persistence (Phase 2) and follow-up period up to 96 weeks. In phase 1 participants will use the DHFS with close follow-up incorporating visits with directly observed ingestions. In Phase 2 the participants utilize the DHFS in their natural setting with sporadic study visits until 12 weeks. Eligible HIV seronegative participants will receive an ingestible sensor enabled oral antiretroviral (IS-ARV) of TDF/FTC (Truvada®). The study will be conducted at the UCSD AVRC. Participants will be recruited from UCSD AVRC, UCSD Owen Clinic, related or affiliated UCSD primary care programs or community primary care clinics. Following the 12 week intervention participants will undergo HIV testing and continuation on HIV PrEP and followed for up to 96 weeks. The primary outcome will be an accurate measure of adherence i.e. the number of doses of selected IS-ARVs ingested, as captured by the DHFS, over the number of doses prescribed, adjusted for positive detection accuracy (PDA), defined as the percentage of detected sensors that have been administered under direct observation.The investigators will also assess the acceptability and feasibility of longitudinal monitoring in real time of the ingestion rate utilizing the DHFS. In addition the investigators will evaluate the ability of the DHFS to identify participants whose longitudinal medication taking and timing patterns in the first 12 weeks of ARV treatment puts them at risk for HIV infection as far out as 96 weeks from start of treatment.

Pharmacokinetic (PK) Substudy

• To obtain TDF/FTC serum levels data comparing co-encapsulated IS-Truvada formulation to native Truvada® as supplemental information to dissolution studies.

A subset of 12 participants prescribed IS-Truvada®:(tenofovir disoproxil fumarate/emtiritabine) for PrEP will be enrolled in a PK sub-study to provide supplementary data to dissolution studies conducted by Gilead Sciences on the co-encapsulated IS-Truvada formulation. On Day 14 of treatment, when drug concentrations are expected to be close to steady state, sub-study participants will have a PK profile for Tenofovir and Emtricitabine obtained over a single dosing interval (at time 0 (pre-dose Ctrough), 2, 4, 6, 8 and 24 hours). Participants will be seen at the AVRC in a fasting state prior to taking their dose of IS-Truvada® and will remain fasting for 2 hours after the observed ingestion. The time and date of the previous doses of IS-Truvada® will be recorded by and available from the DHFS prior to initiating the PK procedures. The following day, Day 15, the participant will return to the AVRC in a fasting state. The 24 hour plasma sample will be drawn. Participants will then receive an observed dose of native Truvada. Participants will remain fasting for 2 hours after the observed ingestion and will have plasma samples drawn at 2, and 4 hours after ingestion.

Samples will be analyzed for tenofovir and emtricitabine drug concentration levels either individually or in batches at the central specialized laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Adult non-pregnant HIV-seronegative participants who are starting or continuing HIV PrEP with IS-TDF/FTC (Truvada®), who are able to use the DHFS mobile device, and to tolerate a wearable sensor patch
2. Laboratory values obtained by screening laboratories within 14 days of entry:

   * Absolute neutrophil count (ANC) ≥ 1,000/mm3.
   * Hemoglobin ≥ 9.0 g/dL.
   * Platelet count ≥ 75,000/mm3.
   * Aspartate aminotransferase (AST) , Alanine aminotransferase (ALT) , and alkaline phosphatase ≤ 3 x ULN.
   * Estimated Glomerular Filtration Rate (GFR) by Cockcroft-Gault equation of >50 ml/min, if starting treatment with Truvada®(TDF/FTC).
   * HIV Ag/Ab test negative
   * Hepatitis B serology negative
3. Females of childbearing potential must agree to use an acceptable form of contraception throughout the protocol.
4. Basic competency in understanding written and verbal information as it applies to DHFS use. English and Spanish will be used for study documents and communication.
5. Willing to follow all protocol requirements.
6. No symptoms or clinical suspicion of acute HIV infection.

Exclusion Criteria:

1. Female who is pregnant, breast-feeding, or of childbearing potential and declines to use contraception throughout the study period.
2. Use of any of the prohibited medications or other non-informed medications within 30 days of study entry (Day 0).
3. Known allergy/sensitivity to any of the study drugs.
4. Known sensitivity to skin adhesives.
5. Serious medical (serious infection or acute therapy for other medical illness) or psychiatric illness requiring systemic treatment and/or hospitalization until participant either completes therapy or is clinically stable on therapy, in the opinion of the investigators, for at least 30 days prior to study entry (Day 0).
6. Active drug or alcohol use, or dependence, or other conditions that, in the opinion of the site investigators, would significantly interfere with ability to follow to study requirements.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication Taking Adherence | 12 weeks
  Medication taking adherence, defined as the number of doses ingested as captured by the DHFS over the number of doses prescribed, adjusted for Positive Detection Accuracy ( determined by the percentage of PrEP medication ingestion detected by the DHFS administered under witnessed observation).
The system positive detection accuracy (PDA) will be derived | 12 weeks
  2. PDA is determined by the percentage of HIV PrEP ingestion detected by the DHFS administered under witnessed observation, overall for all study subjects. PDA will be based upon proper DHFS use. The PDA will be calculated for a single tablet regimen.

SECONDARY OUTCOMES:
Determine the percentage of participants starting or continuing HIV PrEP who find the DHFS acceptable and easy to use. | 12 weeks
  Acceptability and participant satisfaction with the DHFS will be accessed based on the self-report DHFS User Experience questionnaires which include open ended questions and a detailed exit DHFS User Experience questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sara H Browne, MD MPH, Study Chair — UCSD AntiViral Research Center; Constance A Benson, MD, Study Chair — UCSD AntiViral Research Center
Locations (2):
- United States (2):
  - UCSD AntiViral Research Center, San Diego, California
  - San Ysidro Health, San Diego, California